CLINICAL TRIAL: NCT03188835
Title: Brown Fat Energy Metabolism During Cold Exposure: Effects of Fructose- or Glucose-rich Diet in Healthy Subjects
Brief Title: Effects of Fructose/Glucose-rich Diet on Brown Fat in Healthy Subjects (GB7)
Acronym: GB7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: McMaster University (Other); University of Ottawa (Other)
Responsible Party: Principal Investigator, André Carpentier, tenured professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2017-1459
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Diet; Fluorodeoxyglucose F18; carbon-11 acetate; Electromyography; Calorimetry, Indirect

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Isocaloric Diet (Other): Two weeks of isocaloric diet
  Interventions: Other: cold exposure; Radiation: 18FDG; Radiation: 11C-acetate; Radiation: [3-3H]-glucose; Other: [U-13C]-palmitate; Other: 2H-Glycerol; Device: MRI/MRS; Device: Electromyogram (EMG); Device: DXA; Device: Indirect calorimetry
- Fructose diet (Other): Two weeks of hypercaloric diet supplemented with fructose
  Interventions: Dietary Supplement: Diet; Other: cold exposure; Radiation: 18FDG; Radiation: 11C-acetate; Radiation: [3-3H]-glucose; Other: [U-13C]-palmitate; Other: 2H-Glycerol; Device: MRI/MRS; Device: Electromyogram (EMG); Device: DXA; Device: Indirect calorimetry
- Glucose diet (Other): Two weeks of hypercaloric diet supplemented with glucose
  Interventions: Dietary Supplement: Diet; Other: cold exposure; Radiation: 18FDG; Radiation: 11C-acetate; Radiation: [3-3H]-glucose; Other: [U-13C]-palmitate; Other: 2H-Glycerol; Device: MRI/MRS; Device: Electromyogram (EMG); Device: DXA; Device: Indirect calorimetry

INTERVENTIONS:
Dietary Supplement: Diet — A 2 weeks of hypercaloric diet supplemented with fructose or glucose
  Arms: Fructose diet; Glucose diet
Other: cold exposure — Acute cold exposure using a water-conditioned cooling suit will be applied from time 0 to 180 min. At the same time mean skin temperature will be measured by 11 thermocouples.
Radiation: 18FDG — I.v. injection of 18-fluorodeoxyglucose (18FDG) will be performed, followed by 30 min dynamic and 50 min wholebody PET/CT scanning.
Radiation: 11C-acetate — i.v. injection of 11C-acetate will be performed, followed by 20 min dynamic PET/CT scanning
Radiation: [3-3H]-glucose — i.v. administration of 1.5 uCi/min of [3-3H]-glucose
Other: [U-13C]-palmitate — i.v. administration of 0.08 umol/kg/min of [U-13C]-palmitate
Other: 2H-Glycerol — i.v. administration of 0.05 µmol/kg/min of 2H-glycerol
Device: MRI/MRS — Visceral and cervico-thoracic MRI and MRS acquisition.
Device: Electromyogram (EMG) — Skeletal muscle activity and shivering intensity will be measured by electromyography using surface electrodes
Device: DXA — Lean mass will be determined by dual-energy X-ray absorptiometry
Device: Indirect calorimetry — VCO2 will be measured by indirect calorimetry between 15 and 20 min every hour until time 180.

SUMMARY:
Activating brown and beige adipose tissue (herein described as BAT) has been recently recognized as a potential means to increase energy expenditure and lower blood glucose, however, BAT activity appears to be reduced with obesity, aging or Type 2 Diabetes (T2D). BAT has the unique capability to burn large amounts of sugar and fat and effectively dissipate this energy as heat due to the expression of uncoupling protein 1 (UCP1) which is controlled by a thermogenic gene program of transcription factors, co-activators and protein kinases. Thus, enhancing the thermogenic gene program may be beneficial for treating obesity and T2D. Despite the importance of BAT in regulating metabolism our understanding of the factors which suppress its metabolic activity with obesity, aging and T2D are largely unknown. Recently, it was shown that peripheral serotonin, which is regulated by the tryptophan hydroxylase 1 (Tph1), is a negative regulator of BAT metabolic activity. In addition to serotonin, other studies have indicated that pro-inflammatory stimuli may also inhibit BAT metabolic activity. These data suggest that reduced activation of BAT may be due to increases in peripheral serotonin and inflammation. Importantly, the gut microbiome has recently been recognized as an important regulator of serotonin and inflammatory pathways suggesting the observed effects of the microbiome on obesity, T2D may be mediated in part through reductions in BAT activity.

One mechanism by which the environment may impact BAT activity and the thermogenic gene program over the last 3 decades involves changes in our food supply as result of changes in agricultural production (chlorpyrifos, glyphosphate) and the addition of food additives (fructose). These agents have been reported to alter inflammation, serotonin metabolism and the gut microbiome indicating a potential bimodal (direct and indirect via the microbiome) mechanism by which they may alter the thermogenic gene program and contribute to chronic metabolic disease. Thus, our overarching hypothesis is that environmental agents and additives related to food production may contribute to the reduced metabolic activity of BAT. The objective is to identify and characterize how food production agents and additives reduce the metabolic activity of BAT.

DETAILED DESCRIPTION:
Each subject will follow 3 metabolic studies (A, B and C), each lasting 7.5h which includes a 3h acute cold exposure.

These studies will be almost identical: same perfusion of tracers, same number of Positron Emission Tomography (PET) acquisitions and same number of Magnetic Resonance Imaging (MRI) associated with Magnetic Resonance Spectroscopy (MRS) acquisitions .

The difference will be in the diet ingested by the subjects two weeks before each metabolic study: during protocol A, the subjects will follow an isocaloric diet; during protocol B, the subjects will follow the same isocaloric diet supplemented with a daily beverage containing +25% of energy intake from fructose; and during protocol C, the subjects will follow the same isocaloric diet supplemented with a daily beverage containing +25% of energy intake from glucose.

Stool samples will be collected for each metabolic study for microbiome flora and metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects: subjects with normal glucose tolerance determined according to an oral glucose tolerance test and with a BMI < 27 kg/m2 without first degree of familial history of type 2 diabetes (parents, siblings).

Exclusion Criteria:

1. Plasma triglycerides > 5.0 mmol/L at fasting;
2. More than 2 alcohol consumption per day;
3. More than 1 cigarette per day;
4. History of total cholesterol level > 7 mmol/L, of cardiovascular disease, hypertensive crisis;
5. Treatment with fibrates, thiazolidinedione, insulin, beta-blockers or other drugs with effects on insulin resistance or lipid metabolism (exception for anti-hypertensive drugs, statins or metformin);
6. Presence of a non-controlled thyroid disease, renal or hepatic disease, history of pancreatitis, bleeding diatheses, cardiovascular disease or any other serious medical conditions;
7. History of serious gastrointestinal disorders (malabsorption, peptic ulcer, gastroesophageal reflux having required a surgery, etc.);
8. Presence of a pacemaker;
9. Have undergone of PET study or CT scan in the past year;
10. Chronic administration of any medication;

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Microbiome flora | 4 months
  assessed from stool samples
Microbiome metabolites | 4 months
  assessed from stool samples
BAT oxidative metabolism | 4 months
  will be determined using i.v. injection of 11C-acetate during dynamic PET/CT scanning
BAT triglyceride content | 4 months
  will be determined by radiodensity or MRS

SECONDARY OUTCOMES:
BAT blood flow | 4 months
  will be determined using i.v. injection of 11C-acetate during dynamic PET/CT scanning
BAT net glucose uptake | 4 months
  will be assessed using i.v. injection of 18FDG with sequential dynamic PET/CT scanning.
Whole-body glucose partitioning | 4 months
  will be assessed using i.v. injection of 18FDG with static PET/CT scanning
BAT volume of metabolic activity | 4 months
  will be determined using a total body CT (16 mA) followed by a PET acquisition
metabolites appearance rate | 12 months
  will be determined by perfusion of stable isotope tracers
energy metabolism (whole body production) | 4 months
  by indirect calorimetry
hormonal responses | 12 months
  analysed by colorimetric and Elisa tests

CONTACTS AND LOCATIONS:
Overall Officials: André C. Carpentier, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche du CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Richard G, Blondin DP, Syed SA, Rossi L, Fontes ME, Fortin M, Phoenix S, Frisch F, Dubreuil S, Guerin B, Turcotte EE, Lepage M, Surette MG, Schertzer JD, Steinberg GR, Morrison KM, Carpentier AC. High-fructose feeding suppresses cold-stimulated brown adipose tissue glucose uptake independently of changes in thermogenesis and the gut microbiome. Cell Rep Med. 2022 Sep 20;3(9):100742. doi: 10.1016/j.xcrm.2022.100742. PMID 36130480
- See also: High-fructose feeding suppresses cold-stimulated brown adipose tissue glucose uptake independently of changes in thermogenesis and the gut microbiome — https://pubmed.ncbi.nlm.nih.gov/36130480/
- See also: Human brown adipose tissue is not enough to combat cardiometabolic diseases — https://www.jci.org/articles/view/175288